CLINICAL TRIAL: NCT06490679
Title: Evaluation Of Nonsurgical Treatment Of Deep Periodontal Pockets (7-10mm) Using AIRFLOW® Prophylaxis Master Device With Erythritol Powder vs Conventional Instrumentation: A Randomized Controlled Clinical Trial
Brief Title: Evaluation Of Nonsurgical Treatment Of Deep Periodontal Pockets (7-10mm) Using AIRFLOW® Prophylaxis Master Device With Erythritol Powder vs Conventional Instrumentation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammad Alaa Mahmoud Aldawod, Principal Investigator Mohammad Aldawod, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201123 PER 3.3.2
Record Dates: First submitted 2024-06-29; First posted 2024-07-08 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Periodontal Pocket; Periodontitis; Gingival Diseases; Gingival Bleeding
Keywords: Air Abrasive; Erythritol
MeSH Terms: conditions — Periodontal Pocket; Periodontitis; Gingival Diseases; Gingival Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand and ultrasonic scalers and curettes (Experimental): Hand and ultrasonic scalers and curettes will be used for supra- and subgingival instrumentation.
  Interventions: Procedure: Hand and ultrasonic scalers and curettes
- Electro Medical Systems AIRFLOW® Prophylaxis Master Device With Erythritol Powder (Active Comparator): Prophylaxis Master Device With Erythritol Powder An erythritol powder will be used by Electro Medical Systems AIRFLOW® Prophylaxis Master Device.
  Interventions: Device: Electro Medical Systems AIRFLOW® Prophylaxis Master Device

INTERVENTIONS:
Procedure: Hand and ultrasonic scalers and curettes — Combination of ultrasonic and hand instrumentation only. Pockets ≥7 mm will be subgingivally debrided using the piezo device according to manufacturer's instructions, and hand curettes will be used until the operator considers the surfaces to be sufficiently clean and free of deposits.
  Arms: Hand and ultrasonic scalers and curettes
Device: Electro Medical Systems AIRFLOW® Prophylaxis Master Device — (a) Disclosure of biofilm with erythrosine, (b) Removal of supragingival and subgingival (up to 10 mm) biofilm and stains with the use of AIRFLOW® Master Piezon® with AIRFLOW® PLUS powder (EMS-Dental, Nyon Switzerland).
  (c) Supra- and sub-gingival debridement by using the AIRFLOW® Master Piezon® device with Piezon NO PAIN® (EMS-Dental) technology.
  Arms: Electro Medical Systems AIRFLOW® Prophylaxis Master Device With Erythritol Powder

SUMMARY:
Periodontitis is a chronic condition associated with the inflammatory destruction of the periodontal tissues ultimately leading to tooth loss. Clinically, it is identified by key features such as clinical attachment loss (CAL), bleeding upon probing (BOP), and an increase in probing pocket depth (PPD), and/or gingival recession. Periodontitis is mediated by polymicrobial dysbiosis with keystone pathogens affecting the virulence of the entire biofilm community. The removal of this biofilm and its retention factors is the ultimate goal of clinical treatment and oral measures applied. The elimination of the biofilm has traditionally been achieved with the use of either hand instruments or power driven devices. Promoting periodontal health or diminishing bacterial presence and calculus buildup on teeth can be accomplished with the same efficacy whether using manual scalers and curettes or ultrasonic scaling instruments. Both hand and ultrasonic instruments are characterized by being time- consuming and requiring technical skill, often causing patient discomfort and post-treatment pain, including hypersensitivity resulting from the loss of hard tissue when scaling the tooth surface. Ultrasonic instruments tend to leave a rougher surface behind compared to hand instruments. While effective the current techniques all have their disadvantages. The aim of this study is to evaluate changes in probing depth clinically, Bleeding on probing, Clinical attachment level, Plaque index, Calculus index, Patient pain/discomfort, Patient satisfaction, Cost effectiveness, Treatment time and Number of pockets closed after using AIRFLOW® Prophylaxis Master device with erythritol powder.

DETAILED DESCRIPTION:
Patients will be selected from the outpatient clinic of the Oral Medicine and Periodontology Department, Faculty of Dentistry-Cairo University

* Screening of patients will continue until the target sample is achieved. (Consecutive sampling)
* Identifying and recruiting potential subjects will be achieved through patient database.

Preoperative evaluation:

- Clinical examination Each patient will be examined to confirm that he/she met the eligibility criteria.

Age, gender and smoking status will be collected at baseline, along with a complete periodontal charting including 6-point pocket probing depth (PPD), clinical attachment level (CAL), plaque index (PI) according to a modified O'Leary index (O'Leary et al. 1972) measured on 6 surfaces per tooth (distobuccal, buccal, mesiobuccal, distolingual, lingual and mesiolingual), Calculus index according to (Ramfjord SP. 1967).

Periapical x-rays will be taken to confirm the diagnosis of periodontitis.

* Clinical photographs Clinical photographs will be taken at baseline, immediately after treatment and 6 months after treatment.
* Radiographic examination Periapicals radiographs will be taken at the site of interest at baseline and after 3 and 6 months.
* Surgical procedure.

Test sites:

1. Disclosure of biofilm with erythrosine,
2. Removal of supragingival and subgingival (up to 4 mm) biofilm and stains with the use of AIRFLOW® Master Piezon® with AIRFLOW® PLUS powder (EMS- Dental, Nyon Switzerland).
3. Supra- and sub- gingival debridement by using the AIRFLOW® Master Piezon® device with Piezon NO PAIN® (EMS-Dental) technology.

Controls will receive conventional treatment with the combination of ultrasonic and hand instrumentation only. Pockets ≥4 mm will be subgingivally debrided using the piezo device according to manufacturer's instructions, and hand curettes will be used until the operator considers the surfaces to be sufficiently clean and free of deposits.

- Postoperative: At the end of the session, the patients will receive oral hygiene instructions on manual toothbrushing and the use of interdental cleaning devices.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients.
* Patients with an age range between 16 to 80 years.
* Patients have a minimum of 20 teeth.
* Periodontitis patients with at least one residual pocket with a probing depth ranging from 7 to 10 mm.
* Cooperative patients able and willing to come for follow up appointments.

Exclusion Criteria:

* Pregnant and lactation females.
* Patients reporting systemic conditions (eg: diabetes).
* Patients with severe or unstable upper respiratory tract infections, chronic bronchitis/asthma.
* Patients with severe inflammation and/or osteonecrosis.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in probing pocket depth | PPD will be taken at baseline, 1 month, 3 months and 6months after the intervention during the follow-up period and will be done by a single calibrated examiner.
  The PPD will be clinically measured by using UNC 15 periodontal probe from the gingival margin to the depth of the pocket.

SECONDARY OUTCOMES:
Bleeding On Probing | BoP will be taken at baseline, 1 month, 3 months and 6months after the intervention during the follow-up period and will be done by a single calibrated examiner.
  The BoP will be clinically measured by using UNC 15 periodontal probe from the CEJ to the gingival margin.
Clinical Attachment Level | CAL gain will be taken at baseline, 3 months and 6 months after the intervention during the follow-up period and will be done by a single calibrated examiner.
  The CAL will be clinically measured using UNC 15 periodontal probe from the cemento-enamel junction (CEJ) to the depth of defect.
Plaque index | PI will be measured baseline, 1 month, 3 months and 6 months after the intervention during the follow-up period and will be done by a single calibrated examiner
  The PI will be evaluated by using modified O'Leary index teeth are stained with a disclosing solution, presence of plaque is scored on a dichotomous variable and the final score per individual is the sum of the plaque scores divided by the number of surfaces examined.
Calculus index | CI will be taken at baseline, 1 month, 3 months and 6months after the intervention during the follow-up period and will be done by a single calibrated examiner.
  0 =absence of calculus
  1. =supragingival calculus extending only slightly below the free gingival margin (not more than 1 mm.)
  2. = moderate amount of supra and subgingival calculus or subgingival calculus alone
  3. = an abundance of supra and subgingival calculus
Patient pain/discomfort | Postoperative Pain will be measured after the surgical procedure and 1 month, 3 months and 6 months after the intervention
  Postoperative Pain will be measured by using Visual Analogue Score (VAS Score), Minimum 0 = No pain, Maximum 10 = Worst Pain possible
Patient satisfaction | Patient satisfaction will be measured after the surgical procedure and 1 month, 3 months and 6 months after the intervention
  Patient satisfaction will be measured using a survey.
Cost effectiveness | At Baseline and 6 months post-op
  Ratio of cost of treatment and time of procedure against the gained clinical benefit
Treatment time | Up to 6 months
  Time from picking-up the handpiece from the instrument holder to put the handpiece back.
Number of healed pockets | 6 months post-op
  Pocket depth of <3.5 mm clinically measured by using UNC 15 periodontal probe from the gingival margin to the depth of the pocket.

CONTACTS AND LOCATIONS:
Overall Officials: Hani El-Nahas, Professor, Study Director — Cairo University; Omnia Tawfik, Lecturer, Study Chair — Cairo University; Mohammad Aldawod, Bachelor, Principal Investigator — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt